CLINICAL TRIAL: NCT00216112
Title: Imatinib Mesylate (Gleevec®, STI571) in Combination With Docetaxel (Taxotere) for the Treatment of Advanced, Platinum-Refractory Ovarian Cancer and Primary Peritoneal Carcinomatosis: Hoosier Oncology Group GYN03-62
Brief Title: Imatinib Mesylate in Combination With Docetaxel for Advanced, Platinum-Refractory Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniela Matei, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Sanofi (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Daniela Matei, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GYN 03-62
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): Imatinib Mesylate + Docetaxel
  Interventions: Drug: Imatinib Mesylate; Drug: Docetaxel

INTERVENTIONS:
Drug: Imatinib Mesylate — Imatinib mesylate 600 mg po qd
Drug: Docetaxel — Docetaxel 30 mg/m2 (4 of 6 weeks); 1 cycle = 6 weeks

SUMMARY:
Imatinib mesylate is an inhibitor of the receptor tyrosine kinases for platelet-derived growth factor (PDGF) and stem cell factor (SCF), c-Kit, and inhibits PDGF- and SCF-mediated cellular events. Docetaxel promotes cell growth arrest by inhibiting the deassembly of tubulin and by promoting at the same time microtubule assembly. Docetaxel has single agent activity in ovarian cancer with response rates of 30-40% in the platinum refractory setting. The combination of imatinib mesylate and docetaxel has potential synergistic effects, based on previous reports showing synergy in-vitro and in-vivo between PDGFR inhibitors or PI3K inhibitors and taxane chemotherapy.

This trial will investigate the efficacy the combination of imatinib mesylate and docetaxel in treating patients with advanced, platinum-refractory ovarian cancer and primary peritoneal carcinomatosis.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Submit tumor and serum samples for central review

* Imatinib 600 mg (orally qd);
* Docetaxel 30mg/m2 (4 of 6 weeks);1 cycle = 6 weeks
* Evaluate every other cycle

Each cycle will begin only when the granulocyte count is > 1,500/mm3 and the platelet count is > 100,000/mm3 and any other treatment-related toxicities are < grade 1. If the toxicity is not resolved to grade 0 or 1 after three weeks, the patient will be withdrawn from the study. For days 8, 15, and 22 patients must have an absolute neutrophil count > 1,000/mm3 or greater and platelet count > 75,000/mm3. Imatinib mesylate can be administered if platelets >20,000 and ANC >500.

ECOG performance status 0 or 1

Hematopoietic:·

* ANC > 1,500/mm3·
* Platelets > 100,000 mm3·
* Hgb > 8g/dl

Hepatic:·

* Albumin>3gm/dL·
* Total bilirubin < ULN·
* Maximum Alk Phos: >2.5x but < 5x ULN

Renal:·

* Creatinine < 1.5 x ULN·(by Cockroft and Gault)

Cardiovascular:·

* No grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months prior to beginning protocol therapy)

Pulmonary:·

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer·
* Immunohistochemical documentation of c-Kit or PDGFR expression by tumor
* At least one measurable site of disease as defined by RECIST or evidence of disease progression by CA125 measurement
* Platinum-refractory or platinum-resistant

Exclusion Criteria:

* No prior exposure to imatinib (Gleevec®) as single agent or in combination
* No chemotherapy within 28 days (42 days for nitrosourea or mitomycin-C) prior to being registered to protocol therapy.
* No prior radiotherapy to ³ 25 % of the bone marrow
* No known brain metastases.
* Negative pregnancy test
* No current breastfeeding
* No investigational agents within 28 days prior to protocol therapy
* No prior malignancy in the past 5 years unless the other primary malignancy is not currently clinically significant, nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ
* No severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
* No known diagnosis of human immunodeficiency virus (HIV) infection.
* No major surgery within 28 days prior to being registered to protocol therapy.
* No refractory ascites requiring drainage more frequently than once a month
* No presence of clinically significant small bowel obstruction
* No prior exposure to docetaxel (exposure to paclitaxel is allowed)
* No parenteral nutrition within 28 days prior to being registered to protocol therapy.
* No concomitant treatment with potent CYP 3A4 inhibitors (i.e., ketoconazole) is permitted during therapy on this protocol.
* No therapeutic anticoagulation with warfarin while on study (use of low molecular weight heparin is allowed, if necessary).
* No peripheral neuropathy > grade 1
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* No serious concomitant systemic disorders incompatible with the study
* No prior malignancies with the exception of curatively treated basal or squamous carcinoma of the skin, carcinoma in-situ of the cervix, or any other cancer for which the patient has been disease-free for < 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-12; Primary Completion 2005-10 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
· To determine response rate (CR, PR and SD) of patients with advanced, platinum-refractory ovarian cancer, whose tumors over-express PDGFR or c-kit receiving imatinib mesylate in combination with docetaxel. | 24 months

SECONDARY OUTCOMES:
· To assess the safety and tolerability of imatinib mesylate in combination with docetaxel in patients with advanced, platinum-refractory ovarian cancer, whose tumors over-express PDGFR or c-kit. | 24 months
· To determine progression free survival and overall survival in patients with advanced, platinum-refractory ovarian cancer, whose tumors over-express PDGFR or c-kit, receiving imatinib mesylate in combination with docetaxel. | 24 months
· To determine whether basal level of Akt expression or Akt activation (phospho-Akt) in ovarian tumors impacts response to treatment with imatinib and docetaxel. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (9):
- United States (9):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - AP&S Clinic, Terre Haute, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matei D, Emerson RE, Schilder J, Menning N, Baldridge LA, Johnson CS, Breen T, McClean J, Stephens D, Whalen C, Sutton G. Imatinib mesylate in combination with docetaxel for the treatment of patients with advanced, platinum-resistant ovarian cancer and primary peritoneal carcinomatosis : a Hoosier Oncology Group trial. Cancer. 2008 Aug 15;113(4):723-32. doi: 10.1002/cncr.23605. PMID 18618737
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/